CLINICAL TRIAL: NCT00389155
Title: A Multicenter, Randomized Double-Blind Phase II/III Study in the First-Line Treatment of Advanced Transitional Cell Carcinoma (TCC) of the Urothelium Comparing Vinflunine/Gemcitabine to Placebo/Gemcitabine in Patients Who Are Ineligible to Receive Cisplatin-Based Therapy
Brief Title: First-Line Treatment of Advanced Bladder Cancer Randomized vs. Gemcitabine ± Vinflunine in Patients Ineligible to Receive Cisplatin-Based Therapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CA183-002
Record Dates: First submitted 2006-10-17; First posted 2006-10-18 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-11

CONDITIONS: Bladder Cancer; Transitional Cell Carcinoma; Metastasis
Keywords: Advanced or metastatic transitional cell carcinoma of the urothelium
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell; Neoplasm Metastasis | interventions — vinflunine; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vinflunine and gemcitabine (Experimental): solution for injection, IV, vinflunine: 280/320 mg/m2 + gemcitabine: 1000 mg/m2, every 3 wks, variable duration
  Interventions: Drug: Vinflunine; Drug: Gemcitabine
- placebo and gemcitabine (Placebo Comparator): solution for injection, IV, placebo + gemcitabine, 1000 mg/m2, every 3 wks, variable duration
  Interventions: Drug: Gemcitabine; Other: Placebo

INTERVENTIONS:
Drug: Vinflunine — solution for injection, IV, vinflunine: 280/320 mg/m2 + gemcitabine: 1000 mg/m2, every 3 wks, variable duration
  Arms: vinflunine and gemcitabine
Drug: Gemcitabine — solution for injection, IV, placebo + gemcitabine, 1000 mg/m2, every 3 wks, variable duration
Other: Placebo
  Arms: placebo and gemcitabine

SUMMARY:
The purpose of this study is to test an investigational drug, vinflunine (BMS-710485), in combination with gemcitabine in patients with Transitional Cell Carcinoma who cannot be treated with cisplatin. This study will help to determine whether vinflunine in combination with gemcitabine will extend the time period until further growth of the tumor more than gemcitabine alone.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of transitional cell carcinoma of the urothelium that is locally advanced or metastatic
* Ineligible for cisplatin-based therapy because of at least one of the following two medical conditions:

  * Calculated creatinine clearance ≤60 mL/min: OR
  * New York Heart Association Classification Stage III-IV Congestive Heart Failure
* Measurable disease documented by imaging with at least one uni-dimensional lesion
* Adequate performance status (ECOG 0, 1, or 2)
* Men and women ≥18 years of age

Exclusion Criteria:

* Patients in whom radiation or surgery is indicated
* Current neuropathy ≥ CTCAE grade 3
* Prior radiation to ≥ 30% of bone marrow
* Inadequate renal function: serum creatinine clearance ≤ 20 mL/min
* Prior allergy to any vinca alkaloid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Median Progression-free Survival (PFS) as Defined by Response Evaluation Criteria in Solid Tumors (RECIST) Criteria in Participants With Advanced Transitional Cell Carcinoma (TCC) of the Urothelium | Until tumor progression, unacceptable toxicity, withdrawal of patient consent, or discontinuation by investigator decision
  PFS survival is defined as the time between randomization and the date of progression or death, whichever occurs first, before or after treatment discontinuation. For those still on study and those who remain alive and have not progressed after treatment discontinuation, PFS will be censored on the date of the last tumor assessment.

SECONDARY OUTCOMES:
Tumor Response Rate in Participants With A Best Response of Complete (CR) or Partial (PR) as Defined by RECIST criteria | Until tumor progression, unacceptable toxicity, withdrawal of patient consent, or discontinuation by investigator decision
  Tumor response rate is defined as the number of participants in that arm whose best response is PR or CR, divided by the total number of randomized participants in the arm.
Overall Survival of Participants With TCC of the Urothelium | Until tumor progression, unacceptable toxicity, withdrawal of patient consent, or discontinuation by investigator decision
  Survival duration is defined as the time (in months) from randomization until death. For those participants who have not died, survival duration will be censored at the last date the participant was known to be alive.
Disease Control Rate in Participants With Best Response of CR, PR, or Stable Disease (SD) | Until tumor progression, unacceptable toxicity, withdrawal of patient consent, or discontinuation by investigator decision
  Disease control rate is defined as the number of participants in that arm whose best response is PR, CR, or SD, divided by the total number of randomized participants in the treatment arm.
Duration of Response in Participants With Best Response of CR or PR | Until tumor progression, unacceptable toxicity, withdrawal of patient consent, or discontinuation by investigator decision
  Duration of response is computed for participants with best response of CR or PR; the duration is measured from the time measurement criteria are met for CR or PR, whichever is recorded first, until the date of documented progressive disease or death. Participants who neither relapse nor die will be censored on the date of their last tumor assessment.
Number of Participants With Outcome of Death, Serious Adverse Events (SAEs), Adverse Events (AEs) and AEs Leading to Discontinuation | Until tumor progression, unacceptable toxicity, withdrawal of patient consent, or discontinuation by investigator decision
  An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition that does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongs existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in drug dependency or drug abuse, or is an important medical event.
Number of Participants With Serum Chemistry Abnormalities by Worst Common Terminology Criteria (CTC) Grade | Following Day 1 to no longer than 30 days after last dose of study medication
Number of Participants With Abnormal Laboratory Findings by Worst CTC Grade | Following Day 1 to no longer than 30 days after last dose of study medication
Time to Response in Participants With Best Response of CR or PR | Until tumor progression, unacceptable toxicity, withdrawal of patient consent, or discontinuation by investigator decision
  Time to response is defined as the number of months from the first dose of study therapy until measurement criteria are met for PR or CR, whichever is recorded first.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (109):
- United States (64):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Acrc/Arizona Clinical Research Center, Inc., Tucson, Arizona
  - Tower Hematology Oncology Medical Group, Beverly Hills, California
  - Local Institution, Concord, California
  - Glendale Memorial Hospital And Health Center, Glendale, California
  - Moores Ucsd Cancer Center, La Jolla, California
  - North Valley Hematology/Oncology Medical Group, Mission Hills, California
  - Local Institution, Orange, California
  - Stanford University, Stanford, California
  - Local Institution, Newark, Delaware
  - University Of Florida College Of Medicine At Jacksonville, Jacksonville, Florida
  - Local Institution, Jacksonville, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - University Of Miami, Miami, Florida
  - Advanced Medical Specialties, Miami, Florida
  - Medical College Of Georgia, Augusta, Georgia
  - Central Georgia Cancer Care, Pc, Macon, Georgia
  - University Of Chicago, Chicago, Illinois
  - Springfield Clinic, Llp, Springfield, Illinois
  - Michiana Hematology Oncology, P.C., South Bend, Indiana
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Sidney Kimmel Comprehensive Cancer Center At Johns Hopkins, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Mitchell Folbe, Md, Pc, Troy, Michigan
  - Local Institution, Minneapolis, Minnesota
  - Local Institution, Rochester, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - University Of Missouri Healthcare/Ellis Fischel Cancer Ctr, Columbia, Missouri
  - Capital Comprehensive Cancer Care Center, Jefferson City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - Washington University School Of Medicine, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - Hematology Oncology Centers Of The Northern Rockies, Pc, Billings, Montana
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Nevada Cancer Centers, Las Vegas, Nevada
  - The Cancer Center At Hackensack University Medical Center, Hackensack, New Jersey
  - The Mary Imogene Bassett Hospital, Cooperstown, New York
  - Columbia University Medical Center, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - University Of Rochester, Rochester, New York
  - Albert Einstein Cancer Center, The Bronx, New York
  - Carolinas Hematology Oncology Associates, Charlotte, North Carolina
  - Mid Dakota Clinic, Pc, Bismarck, North Dakota
  - Cleveland Clinic, Cleveland, Ohio
  - Mid-Ohio Oncology/Hematology, Inc. Dba, Columbus, Ohio
  - Abramson Cancer Center Of The, Philadelphia, Pennsylvania
  - Guthrie Foundation For Education And Research, Sayre, Pennsylvania
  - Charleston Cancer Center, Charleston, South Carolina
  - Medical University Of South Carolina, Charleston, South Carolina
  - The Jones Clinic, Pc, Germantown, Tennessee
  - The West Clinic, Memphis, Tennessee
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - Lone Star Oncology Consulants, Pa, Austin, Texas
  - Cancer Specialists Of South Texas, Pa, Corpus Christi, Texas
  - The Center For Cancer And Blood Disorders, Fort Worth, Texas
  - University Of Texas Medical Branch Of Galveston, Galveston, Texas
  - South Texas Oncology And Hematology, P.A., San Antonio, Texas
  - Northern Utah Associates, Ogden, Utah
  - Cancer Outreach Associates, Pc, Abingdon, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Univ. Of Washington Medical Ctr., Prostate-Oncology Ctr, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
  - Local Institution, Milwaukee, Wisconsin
- Australia (2):
  - Local Institution, Tweed Heads, New South Wales
  - Local Institution, Adelaide, South Australia
- Belgium (2):
  - Local Institution, Antwerp, Antwerp
  - Local Institution, Edegem
- Canada (4):
  - Local Institution, Moncton, New Brunswick
  - Local Institution, Sydney, Nova Scotia
  - Local Institution, London, Ontario
  - Local Institution, Montreal, Quebec
- Denmark (4):
  - Local Institution, Aarhus
  - Local Institution, Herlev
  - Local Institution, København Ø
  - Local Institution, Odense C
- France (3):
  - Local Institution, Caen
  - Local Institution, Paris
  - Local Institution, Vandœuvre-lès-Nancy
- Local Institution, Athens, Greece
- Local Institution, Jakarta, Indonesia
- Italy (3):
  - Local Institution, Milan
  - Local Institution, Trento
  - Local Institution, Viterbo
- Philippines (4):
  - Local Institution, Cebu
  - Local Institution, Davao City
  - Local Institution, Manila
  - Local Institution, Quezon City
- Poland (6):
  - Local Institution, Bialystok
  - Local Institution, Gdansk
  - Local Institution, Krakow
  - Local Institution, Olsztyn
  - Local Institution, Poznan
  - Local Institution, Warsaw
- Russia (3):
  - Local Institution, Obninsk, Kaluga Oblast
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
- South Korea (2):
  - Local Institution, Seongnam-si, Gyeonggi-do
  - Local Institution, Seoul
- Spain (5):
  - Local Institution, Barcelona
  - Local Institution, Murcia
  - Local Institution, Palma de Mallorca
  - Local Institution, Sabadell (Barcelona)
  - Local Institution, Santander
- Local Institution, Bangkok, Thailand
- United Kingdom (4):
  - Local Institution, Cardiff, Glamorgan
  - Local Institution, Grimsby, Lincolnshire
  - Local Institution, Nottingham, Nottinghamshire
  - Local Institution, Birmingham, West Midlands